CLINICAL TRIAL: NCT04046640
Title: A Study on the Heat Transport Characteristics of Meridian Phenomenon for the Heart and Lung Meridians Based on Patients With Stable Angina Pectoris
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang Chinese Medical University (Other Government)
Collaborators: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other); The First Affiliated Hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Jianqiao Fang, President, Zhejiang Chinese Medical University
Other Study IDs: 2019ZY003-MERIDIAN
Record Dates: First submitted 2019-08-01; First posted 2019-08-06 (Actual); Last update posted 2020-01-22 (Actual); Status verified 2020-01

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: meridians; acupuncture; chronic obstructive pulmonary disease; meridian phenomenon; infrared thermography
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CSAP group: This group will include 40 patients with chronic stable angina pectoris (CSAP).
  Interventions: Device: Infrared thermal imaging
- Healthy group: This group will include 40 healthy volunteers.
  Interventions: Device: Infrared thermal imaging

INTERVENTIONS:
Device: Infrared thermal imaging — Infrared thermal imaging will be adopted to assess the heat transport characteristics of meridian phenomenon for participants in the two groups.
  1. Experimental device: a NEC InfRec R450 infrared thermal imaging camera
  2. Experimental process: The participants will be allowed to stabilize for 15 minutes in a supine position in the experimental room before formal examination They are asked to keep silent, breathe normally and avoid movement of limbs during the whole measuring period. The height and angle of the infrared thermal imaging camera is adjusted so that the measurement sites of the participant's arm is located in the center of the camera screen. The infrared thermal imaging and acupoint temperature will be recorded for 5 minutes.
  3. Measurement sites: Shenmen (HT7) and Shaohai (HT3) of the Heart meridian, Taiyuan(LU9) and Chize (LU5) of the Lung meridian.

SUMMARY:
Although some important progresses were made in the field of the meridian research, no breakthroughs have been achieved. Besides,there are some problems in meridian researches. Particularly, previous research of meridian phenomenon involved lots of subjective elements and outcomes.Researches that use modern scientific techniques to investigate the biological characteristics of meridian phenomenon are urgently needed. Therefore, this study is designed to assess the heat transport characteristics of meridian phenomenon for the Heart and Lung meridians by using infrared thermal imaging. Thus, the biological characteristics of meridian phenomenon could be presented objectively in a scientific methodology.

DETAILED DESCRIPTION:
This study will include 40 patients diagnosed with chronic stable angina pectoris (CSAP) and 40 healthy volunteers. Infrared thermal imaging will be adopted to assess the heat transport characteristics of meridian phenomenon for Heart and Lung meridians in the physiology/pathological state. In addition, by comparing the heat transport characteristics in the acupoints along the Heart and Lung meridians, the relative specificity of the two meridians will also be investigated.

Primary outcomes will be infrared thermal images and acupoint temperature. Furthermore, this study will build standardized techniques and schemes for detecting the heat transport characteristics of meridian phenomenon for Heart and Lung. The results of this study could also provide scientific foundation for traditional meridian theories.

ELIGIBILITY:
Inclusion Criteria:

Inclusion criteria for CSAP

1. Patients should meet the diagnostic criteria of coronary heart disease, which includes the following items: 1)confirmed old myocardial infarction (MI), or a history of percutaneous coronary intervention(PCI), or coronary artery bypass grafting; 2)50% or more luminal stenosis in at least one coronary artery or major branch segment confirmed by coronary angiogram or CT angiography; 3) myocardial ischemia indicted by exercise stress radionuclide myocardial imaging; 4) treadmill exercise testing is positive (for male patients);
2. Patients should meet the diagnostic criteria of CSAP and the Canadian Cardiovascular Society(CCS) classification for CSAP is level II or III;
3. The medical history of angina pectoris ≥3 months, with at least 2 episodes per week in the last month;
4. 35 ≤ age ≤65 years, male or female;
5. Patients have clear consciousness and could communicate with others normally;
6. Patients could understand the full study protocol and have high adherence. Written informed consent is signed by themselves or their lineal kin.

Inclusion criteria for health volunteers

1. Healthy volunteers who could provide a recent (in the past 3 month) medical examination report to confirm they have not any cardiovascular, respiratory, digestive, urinary, hematological, endocrine and neurological disease;
2. 35 ≤ age ≤65 years, male or female;
3. Participants have clear consciousness and could communicate with others normally;
4. Participants could understand the full study protocol and have high adherence .Written informed consent is signed by themselves or their lineal kin.

Exclusion Criteria:

Exclusion criteria for CSAP

1. Patients with acute coronary syndrome (including acute myocardial infarction and unstable angina) and severe arrhythmias (such as severe atrioventricular block, ventricular tachycardia, supraventricular tachycardia, frequent premature beats and premature ventricular contraction);
2. Patients' chest pain is caused by valvular heart disease, hypertrophic cardiomyopathy and dilated cardiomyopathy;
3. Patients' chest pain is caused by non-cardiac disease (such as severe neurosis, climacteric syndrome, cervical spondylosis, and esophageal/pulmonary/chest wall lesions);
4. Patients have concomitant conditions of lung diseases, such as chronic obstructive pulmonary disease (COPD);
5. Patients have serious concomitant conditions and and fail to treat them effectively, such as diseases of the digestive, urinary, respiratory, hematological and nervous system;
6. Patients have mental illness, severe depression, alcohol dependence or history of drug abuse;
7. Pregnant or lactating patients;
8. Patients are participating in other trials.

Exclusion criteria of health volunteers

1. Participants have sudden severe diseases during the trial, such as cardiovascular diseases, liver diseases, kidney diseases, urinary diseases and hematological diseases.
2. Participants have mental illness, severe depression, alcohol dependence or history of drug abuse;
3. Pregnant or lactating participants ;
4. Participants are participating in other trials.

Ages: 35 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: 40 patients with chronic stable angina pectoris (CSAP) and 40 healthy volunteer.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2020-02 (Estimated); Primary Completion 2020-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Infrared thermal images | 5 minutes
  Infrared thermal images could reflect the heat transport characteristics of meridian phenomenon.
Acupoint temperature | 5 minutes
  Acupoint temperature could reflect the heat transport characteristics of meridian phenomenon.

CONTACTS AND LOCATIONS:
Overall Officials: Jianqiao Fang, Principal Investigator — Zhejiang Chinese Medical University
Locations (1):
- the Third affiliated hospital of Zhejiang Chinese Medical university, Hanzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cai W, Chen AW, Ding L, Shen WD. Thermal Effects of Acupuncture by the Infrared Thermography Test in Patients With Tinnitus. J Acupunct Meridian Stud. 2019 Aug;12(4):131-135. doi: 10.1016/j.jams.2019.05.002. Epub 2019 Jun 27. PMID 31254681
- [Background] Alvarez-Prats D, Carvajal-Fernandez O, Valera Garrido F, Pecos-Martin D, Garcia-Godino A, Santafe MM, Medina-Mirapeix F. Acupuncture Points and Perforating Cutaneous Vessels Identified Using Infrared Thermography: A Cross-Sectional Pilot Study. Evid Based Complement Alternat Med. 2019 Mar 21;2019:7126439. doi: 10.1155/2019/7126439. eCollection 2019. PMID 31015854
- [Background] Lin M, Wei H, Zhao L, Zhao J, Cheng K, Deng H, Shen X, Zhang H. [Review on infrared temperature characteristics of acupoints in recent 10 years]. Zhongguo Zhen Jiu. 2017 Apr 12;37(4):453-456. doi: 10.13703/j.0255-2930.2017.04.028. Chinese. PMID 29231602
- [Background] Fu Y, Ni JX, Marmori F, Zhu Q, Tan C, Zhao JP. Infrared thermal imaging-based research on the intermediate structures of the lung and large intestine exterior-interior relationship in asthma patients. Chin J Integr Med. 2016 Nov;22(11):855-860. doi: 10.1007/s11655-016-2102-4. Epub 2016 Jun 9. PMID 27286712
- [Background] de Souza RC, Pansini M, Arruda G, Valente C, Brioschi ML. Laser acupuncture causes thermal changes in small intestine meridian pathway. Lasers Med Sci. 2016 Nov;31(8):1645-1649. doi: 10.1007/s10103-016-2032-6. Epub 2016 Aug 5. PMID 27495129
- [Background] Yang H, Park H, Lim C, Park S, Lee K. Infrared thermal imaging in patients with medial collateral ligament injury of the knee - a retrospective study. J Pharmacopuncture. 2014 Dec;17(4):50-4. doi: 10.3831/KPI.2014.17.036. PMID 25780719
- [Background] Zheng J, Zhao Y, Wang Y, Hu S, Lu P, Shen X. The infrared radiation temperature characteristic of acupoints of mammary gland hyperplasia patients. Evid Based Complement Alternat Med. 2013;2013:567987. doi: 10.1155/2013/567987. Epub 2013 Nov 14. PMID 24327822
- [Background] Kang J, Lee N, Ahn Y, Lee H. Study on improving blood flow with Korean red ginseng substances using digital infrared thermal imaging and Doppler sonography: randomized, double blind, placebo-controlled clinical trial with parallel design. J Tradit Chin Med. 2013 Feb;33(1):39-45. doi: 10.1016/s0254-6272(13)60098-9. PMID 23596810
- [Derived] Jiang Y, Li X, He X, Hu H, Zhang Y, Shao X, Fang J. The specificity for the correlation between viscera and somato in chronic stable angina pectoris patients and healthy controls: An assessor-blinded and comparative trial. PLoS One. 2025 Sep 26;20(9):e0331868. doi: 10.1371/journal.pone.0331868. eCollection 2025. PMID 41004484

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04046640/Prot_SAP_000.pdf
  • Informed Consent Form (2019-03-25): https://cdn.clinicaltrials.gov/large-docs/40/NCT04046640/ICF_001.pdf